CLINICAL TRIAL: NCT01143805
Title: A Phase 1, Open Label, Single Dose, Randomized, Cross Over Study To Estimate The Absolute Oral Bioavailability Of CP-690,550 In Healthy Subjects
Brief Title: A Study To Estimate The Amount Of CP-690,550 (Study Drug) That Is Absorbed Into The Blood Of Healthy Subjects Following Oral Administration Of CP-690,550 In Tablet Form
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3921077
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Absolute Bioavailability; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Tablets; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Tasocitinib 10 mg oral tablet (Experimental)
  Interventions: Drug: Tasocitinib 10 mg oral tablet
- Treatment B: Tasocitinib 10 mg IV Infusion (Experimental)
  Interventions: Drug: Tasocitinib 10 mg IV Infusion

INTERVENTIONS:
Drug: Tasocitinib 10 mg oral tablet — Treatment A: Single-dose of tasocitinib (CP-690,550) (10 mg) in the form of an oral tablet
  Arms: Treatment A: Tasocitinib 10 mg oral tablet
Drug: Tasocitinib 10 mg IV Infusion — Treatment B: Single-dose of tasocitinib (CP-690,550) (10 mg) in the form of a 30 minute intravenous infusion
  Arms: Treatment B: Tasocitinib 10 mg IV Infusion

SUMMARY:
In this study, a 10 mg dose of CP-690,550 will be given to study subjects on two separate occasions by two different routes of administration: One time by mouth in tablet form and one time by vein (intravenous form). The amount of CP-690,550 available in the blood following administration by vein will be measured and is expected to reflect the maximum amount possible for the 10 mg CP-690,550 dose. The amount of CP-690,550 that is achieved in the blood following oral tablet administration will also be measured and compared to that achieved following administration by vein in order to estimate how much of the maximum amount possible is actually absorbed into the blood following administration by mouth as a tablet.

DETAILED DESCRIPTION:
To estimate the absolute bioavailability of a 10 mg oral dose of tasocitinib (CP-690,550) compared to a 10 mg intravenous dose of tasocitinib (CP-690,550) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non childbearing potential)
* Subjects between the ages of 21 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Exclusion Criteria:

* Evidence or history of any clinically significant illness, medical condition, or disease.

  2. Evidence or history of any clinically significant infections within the past 3 months.

  3. Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
AUCinf of tasocitinib (CP 690,550) | PK blood samples out to 12 hours post dose

SECONDARY OUTCOMES:
AUClast, Cmax, Tmax, and t½, CL (IV dose only) and Vss (IV dose only) of tasocitinib (CP 690,550). | PK blood samples out to 12 hours postdose
Safety Laboratory tests: hematology, chemistry, urine testing | Safety Laboratory testing performed out to 2 days post last dose
Vital Signs: Blood pressure, heart rate, oral temperature | Vital signs out to 2 days post last dose
AE Reporting | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921077&StudyName=A%20Study%20To%20Estimate%20The%20Amount%20Of%20CP-690%2C550%20%28Study%20Drug%29%20That%20Is%20Absorbed%20Into%20The%20Blood%20Of%20Healthy%20Subjects%20Following%20Oral%20A